CLINICAL TRIAL: NCT02907359
Title: A Phase 3, Multicenter, Randomized, Open-Label Study of Guadecitabine (SGI-110) Versus Treatment Choice in Adults With Myelodysplastic Syndromes (MDS) or Chronic Myelomonocytic Leukemia (CMML) Previously Treated With Hypomethylating Agents
Brief Title: Guadecitabine (SGI-110) vs Treatment Choice in Adults With MDS or CMML Previously Treated With HMAs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGI-110-07; 2015-005257-12 (EudraCT Number)
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Results first posted 2023-05-18 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Guadecitabine (Experimental): Participants received Guadecitabine 60 mg/m^2, SC, on Days 1-5 of each 28-day cycle for at least 6 cycles in the absence of unacceptable toxicity or disease progression requiring alternative therapy. Participants received Guadecitabine treatment beyond 6 cycles as long as the participant continued to benefit based on investigator judgment and participant response and tolerability (or up to a maximum of 36 cycles).
  Interventions: Drug: Guadecitabine
- Treatment Choice (Active Comparator): Participants received one of the three treatment choice options:
  1. LDAC 20 mg/m^2 SC/IV once daily for 14 days of each 28-day cycles for at least 4 cycles in absence of disease progression or unacceptable toxicity.Participants who were responding or had stable disease were to continue treatment as per standard institutional practice.
  2. Standard IC of a 7+3 regimen:Cytarabine 100-200 mg/m^2/day given as continuous infusion for 7 days and anthracycline(daunorubicin(45-60 mg)/idarubicin(9-12 mg)/mitoxantrone(8-12 mg)/m^2) by IV infusion for 3 days of each 28-day cycles.
  3. BSC as needed during the treatment included,but was not limited to,blood transfusions(RBCs or platelets),growth factors including erythropoiesis stimulating agents,granulocyte stimulating factors,iron chelating therapy,and broad-spectrum antibiotics and/or antifungals.
  Duration for treatment choice was as per locally approved prescribing information and institutional standard practice or up to a maximum 30 cycles.
  Interventions: Other: Treatment Choice

INTERVENTIONS:
Drug: Guadecitabine
  Other Names: SGI-110
  Arms: Guadecitabine
Other: Treatment Choice — * BSC: according to standard/institutional practice; included RBC or platelet transfusions; growth factors, i.e. erythropoiesis stimulating agents, granulocyte stimulating factors, iron chelating therapy; broad spectrum antibiotics and/or antifungals.
  * LDAC: 20 mg/m^2 SC or IV once daily (QD) for 14 days in 28-day cycles. Other schedules were allowed per institutional practice. Treatment for ≥4 cycles absent disease progression/toxicity. BSC per institutional/standard practice.
  * Standard Intensive Chemotherapy: recommended regimen of 7+3 was given as cytarabine 100-200 mg/m^2/day continuous infusion for 7 days and an anthracycline for 3 days. Anthracyclines per institutional practice included daunorubicin (45-60 mg/m^2/day) or idarubicin (9-12 mg/m^2/day) or mitoxantrone (8-12 mg/m^2/day) by IV infusion. Participants with complete or partial response after IC induction received ≥1 additional cycles with reduced cytotoxic doses then BSC per standard /institutional practice.
  Arms: Treatment Choice

SUMMARY:
A Phase 3, randomized, open-label, parallel-group, multicenter study designed to evaluate the efficacy and safety of guadecitabine in participants with MDS or CMML who failed or relapsed after adequate prior treatment with azacitidine, decitabine, or both. This global study will be conducted in approximately 15 countries. Approximately 408 participants from approximately 100 study centers will be randomly assigned in a 2:1 ratio to either guadecitabine (approximately 272 participants) or Treatment Choice (approximately 136 participants). The study consists of a 21-day screening period, a treatment period, a safety follow-up visit, and a long-term follow-up period. The study is expected to last more than 2 years, and the duration of individual participant participation will vary. Participants may continue to receive treatment for as long as they continue to benefit.

DETAILED DESCRIPTION:
Multicenter, randomized, open-label, parallel-group study of guadecitabine vs Treatment Choice (TC). Approximately 408 participants will be randomly assigned 2:1 to either guadecitabine or TC.

* Guadecitabine: approximately 272 participants.
* TC: approximately 136 participants.

Before randomization, the investigator will assign each participant to one of the following TC options:

* Low dose cytarabine (LDAC).
* Standard Intensive Chemotherapy (IC) of a 7+3 regimen.
* Best Supportive Care (BSC) only. BSC will be provided to all participants as per standard and institutional practice. Participants randomized to TC will not be allowed to cross over to guadecitabine. Data will be reviewed by an independent Data Monitoring Committee at regular intervals, primarily to evaluate safety during study conduct. Randomization will be stratified by disease category (MDS vs CMML), bone marrow (BM) blasts (BM blasts >10% vs BM blasts ≤10%), TC option (LDAC vs IC vs BSC), and study center region.

Guadecitabine: 60 milligrams per square meter (mg/m^2) given subcutaneously (SC) daily on Days 1-5 in 28-day cycles (delayed as needed to allow blood count recovery). Treatment should be given for at least 6 total cycles in the absence of unacceptable toxicity or disease progression requiring alternative therapy. Beyond 6 cycles, treatment should continue as long as the participant continues to benefit. BSC should be given according to standard and institutional practice.

Treatment Choice (TC): Before randomization, the investigator will assign each participant to one of the following TC options:

* Low dose cytarabine (LDAC) given as 20 mg/m^2 SC or intravenously (IV) once daily for 14 days in 28-day cycles (delayed as needed to allow blood count recovery). Treatment should be given for at least 4 cycles in the absence of disease progression or unacceptable toxicity.
* Standard Intensive Chemotherapy (IC) of a 7+3 regimen: given as cytarabine 100-200 mg/m^2/day given as continuous infusion for 7 days and an anthracycline given as per institutional standard practice such as daunorubicin (45-60 mg/m^2/day), or idarubicin (9-12 mg/m^2/day), or mitoxantrone (8-12 mg/m^2/day) by intravenous infusion for 3 days.
* Best Supportive Care (BSC) only: given according to standard and institutional practice. BSC includes, but is not limited to blood transfusions (Red blood cells [RBCs] or platelets), growth factors including erythropoiesis stimulating agents (ESA), granulocyte stimulating factors (GSFs), iron chelating therapy, and broad-spectrum antibiotics and/or antifungals.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥18 years of age who are able to understand and comply with study procedures and provide written informed consent before any study-specific procedure.
* Cytologically or histologically confirmed diagnosis of MDS or CMML according to the 2008 World Health Organization (WHO) classification.
* Performance status (ECOG) of 0-2.
* Previously treated MDS or CMML, defined as prior treatment with at least one hypomethylating agent (HMA; azacitidine and/or decitabine) for intermediate or high risk MDS or CMML whose disease progressed or relapsed as follows:

  1. Participant received HMA for at least 6 cycles and was still transfusion dependent.
  2. Participant received HMA for at least 2 complete cycles and had disease progression prior to Cycle 6 defined as

  i. ≥50% increase in bone marrow blasts from pre-HMA-treatment levels or from nadir post-HMA-treatment levels to >5% (for participants with pretreatment or nadir blasts ≤5%) or to >10% (for participants with pretreatment or nadir blasts >5%), and/or ii. Transfusion dependent and ≥2 gram/deciliter (g/dL) reduction of Hgb from pre-HMA-treatment levels.

Other prior treatments for MDS such as lenalidomide, cytarabine, intensive chemotherapy, hydroxyurea, erythropoietin and other growth factors, or hematopoietic cell transplant (HCT) are allowed.

* Participants must have either:

  1. Bone marrow blasts >5% at randomization, OR
  2. Transfusion dependence, defined as having had transfusion (in the setting of active disease) of 2 or more units of RBC or platelets within 8 weeks prior to randomization.
* Creatinine clearance or glomerular filtration rate ≥30 milliliter/minute (mL/min) estimated by the Cockroft-Gault (C-G) or other medically acceptable formulas such as MDRD (Modification of Diet in Renal Disease) or CKD-EPI (the Chronic Kidney Disease Epidemiology Collaboration).
* Women of childbearing potential must not be pregnant or breastfeeding and must have a negative pregnancy test at screening. Women of childbearing potential and men with female partners of childbearing potential must agree to practice 2 highly effective contraceptive measures of birth control and must agree not to become pregnant or father a child (a) while receiving treatment with guadecitabine and for at least 3 months after completing treatment and (b) while receiving treatment with LDAC or IC and for at least 6 months after completing treatment or for the duration specified in local prescribing information, whichever is longer.

Exclusion Criteria:

* Participants who have been diagnosed as having AML with peripheral blood or bone marrow blasts of ≥20%.
* Participants who may still be sensitive to repeated treatment with decitabine or azacitidine such as participants who had response to prior decitabine or azacitidine treatment, but relapsed >6 months after stopping treatment with these agents.
* Prior treatment with guadecitabine.
* Hypersensitivity to decitabine, guadecitabine, or any of their excipients.
* Second malignancy currently requiring active therapy, except breast or prostate cancer stable on or responding to endocrine therapy.
* Treated with any investigational drug within 2 weeks of the first dose of study treatment.
* Total serum bilirubin >2.5 × upper limit of normal (ULN) (except for participants with Gilbert's Syndrome for whom direct bilirubin is <2.5×ULN), or liver cirrhosis or chronic liver disease Child-Pugh Class B or C.
* Known active HIV, HBV, or HCV infection. Inactive hepatitis carrier status or low viral hepatitis titer on antivirals is allowed.
* Known significant mental illness or other condition such as active alcohol or other substance abuse or addiction that, in the opinion of the investigator, predisposes the participant to high risk of noncompliance with the protocol.
* Refractory congestive heart failure unresponsive to medical treatment, active infection resistant to all antibiotics, or advanced non-MDS associated pulmonary disease requiring >2 liters per minute oxygen.
* Life expectancy of less than one month
* Participants with TP53 mutations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Sano, MD, PhD, Study Director — Astex Pharmaceuticals, Inc.
Locations (112):
- United States (22):
  - City of Hope, Duarte, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Cancer Specialists of North Florida, Fleming Island, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - North Shore Medical Center, Evanston, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke Cancer Center, Durham, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Greenville, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University Mary Babb Randolph Cancer Center, Morgantown, West Virginia
- Belgium (3):
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende, Bruges
  - Grand Hôpital de Charleroi - Notre Dame, Charleroi
- Canada (9):
  - Tom Baker Cancer Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Burnaby Hospital, Burnaby
  - Moncton Hospital, Moncton
  - Maisonneuve-Rosemont Hôpital Service d'Hematologie et d'Oncologie Medicale, Montreal
  - Saskatchewan Cancer Agency, Regina
- Czechia (5):
  - Fakultní nemocnice Brno, Brno
  - Fakultni Nemocnice Hradec Králové, Hradec Králové
  - Fakultní nemocnice Ostrava, Ostrava
  - Fakultní Nemocnice Královské Vinohrady, Prague
  - Onkologická klinika Všeobecná fakultní nemocnice v Praze a 1, Prague
- Denmark (4):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- France (8):
  - Centre Hospitalier Universitaire, La Tronche
  - Hôpital Dupuytren, Limoges
  - GHR Mulhouse Sud-Alsace, Mulhouse
  - Hôpital Hôtel-Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Germany (5):
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Marien Hospital Düsseldorf, Düsseldorf
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum Ulm, Ulm
- Italy (8):
  - Azienda Ospedaliera SS. Antonio E. Biagio E. Cesare Arrigo di Alessandria, Alessandria
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - AORN A. Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria-Maggiore della Carità di Novara, Novara
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - Ospedale S. Eugenio, Roma
- Japan (22):
  - NHO Nagoya Medical Center, Nagoya, Aichi-ken
  - Narita Red Cross Hospital, Narita, Chiba
  - University of Fukui Hospital, Yoshida, Fukui
  - Chugoku Central Hospital, Fukuyama-shi, Hiroshima
  - Tokai University Hospital, Isehara, Kanagawa
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Yokohama Municipal Citizen's Hospital, Yokohama, Kanagawa
  - Nagasaki University Hospital, Nagasaki, Nagasaki-shi
  - Kansai Medical University Hirakata, Hirakata, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Nippon Medical School Hospital, Bunkyō-Ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto, Tokyo
  - NTT Medical Center Tokyo, Shinagawa, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - National Hospital Organization Kyushu, Fukuoka
  - Fukushima Medical University, Fukushima
  - Gifu Municipal Hospital, Gifu
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - University Hospital-Kyoto Prefectural University of Medicine, Kyoto
  - Yamagata University Hospital, Yamagata
- Poland (3):
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- South Korea (6):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (11):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Fundació Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital de León, León
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Östra sjukhuset, Gothenburg
  - Universitetssjukhuset Örebro, Örebro
- United Kingdom (4):
  - Medway NHS Foundation Trust, Gillingham
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 101 investigative sites in the United States, Canada, Spain, Italy, France, Germany, Czech Republic, Denmark, Poland, Belgium, Sweden, United Kingdom, Japan, and South Korea from 13 January 2017 to 30 November 2020.
Pre-assignment Details: A total of 417 participants were randomized (277 in Guadecitabine arm group and 140 in Treatment Choice arm group) and 392 received treatment. Of 417 participants, 48 completed the study.
Groups:
- Guadecitabine: Participants received Guadecitabine 60 milligrams per square meter (mg/m^2), subcutaneously (SC), on Days 1-5 of each 28-day cycle for at least 6 cycles in the absence of unacceptable toxicity or disease progression requiring alternative therapy. Participants received Guadecitabine treatment beyond 6 cycles as long as the participant continued to benefit based on investigator judgment and participant response and tolerability (or up to a maximum of 36 cycles).
- Treatment Choice: Participants received one of the three treatment choice options:
  1. Low dose cytarabine (LDAC) 20 mg/m^2 SC or intravenous (IV) once daily for 14 days of each 28-day cycles for at least 4 cycles in the absence of disease progression or unacceptable toxicity. Participants who were responding or had stable disease were to continue treatment as per standard and institutional practice.
  2. Standard Intensive Chemotherapy (IC) of a 7+3 regimen: Cytarabine 100-200 mg/m^2/day given as continuous infusion for 7 days and an anthracycline (daunorubicin (45-60 mg)/idarubicin (9-12 mg)/mitoxantrone (8-12 mg)/m^2) by IV infusion for 3 days of each 28-day cycles.
  3. Best Supportive Care (BSC) as needed during the treatment included, but was not limited to, blood transfusions (Red blood cells [RBCs] or platelets), growth factors including erythropoiesis stimulating agents, granulocyte stimulating factors, iron chelating therapy, and broad-spectrum antibiotics and/or antifungals.
  Duration for treatment choice was as per locally approved prescribing information and institutional standard practice or up to a maximum 30 cycles.
Period: Overall Study
Arm/Group | Guadecitabine | Treatment Choice
Started (The Efficacy Analysis Set included all participants randomly assigned to the study treatment.) | 277 | 140
Safety Analysis Set (The Safety Analysis Set included all participants randomly assigned to study treatment who received any amount of study treatment or any component of a multi-dose study treatment regimen.) | 270 | 122
Completed | 36 | 12
Not Completed | 241 | 128
Not completed — Death | 234 | 117
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Guadecitabine | Treatment Choice | Total
Number analyzed (Participants) | 277 | 140 | 417
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (7) | 73.7 (6.1) | 73.6 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 44 | 127
  Male | 194 | 96 | 290
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 7 | 31
  Not Hispanic or Latino | 225 | 117 | 342
  Unknown or Not Reported | 28 | 16 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 64 | 33 | 97
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  White | 179 | 86 | 265
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 16 | 45

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the number of days from the day the participant was randomized to the date of death due to any cause. Survival time was censored on the last date the participant is known alive with no event of death. OS time will be estimated using the Kaplan-Meier method.
Time Frame: From randomization up to death (up to approximately 38.6 months)
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 277 | 140
days | 277.0 [243.0 to 313.0] | 252.0 [200.0 to 325.0]
Statistical Analysis 1: Comparison: Guadecitabine vs Treatment Choice; Test type: Superiority; p = 0.6063, Stratified Log-rank test — OS between Guadecitabine vs Treatment Choice using stratified log-rank test. Due to pre-specified hierarchical testing plan, other endpoints were not evaluated for statistical significance; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.74 to 1.19]

2. Secondary Outcome: Percentage of Participants With Transfusion Independence for Any 8 Consecutive Weeks
Description: Transfusion independence rate was calculated as the number of participants with neither RBC nor platelet transfusion for any period of 8 weeks after the initiation of treatment (or cycle 1 day 1 { C1D1} visit date for participants randomized to BSC or randomization date for participants not treated) and up to treatment discontinuation (or 180 days for participants discontinuing the treatment within 6 months), while maintaining haemoglobin (Hgb) ≥8 gram per deciliter (g/dL) and platelets ≥20×10^9/liter (L) divided by the total number of participants included in the efficacy analysis. RBC or Platelet transfusion independence rate was defined similarly as above. Percentage of participants are rounded off to the single decimal point.
Time Frame: Up to approximately 46.6 months
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 277 | 140
percentage of participants
  Transfusion Independence Rate (8 weeks) | 15.9 | 15.7
  Platelet Transfusion Independence Rate | 32.1 | 37.9
  RBC Transfusion Independence Rate | 22.4 | 22.0

3. Secondary Outcome: Percentage of Participants With Marrow Complete Response (mCR) Along With Transfusion Independence Rate
Description: mCR was defined as per 2006 Myelodysplastic Syndromes International Council for Harmonisation (MDS IWG) criteria as reduction of bone marrow (BM) blasts to ≤5% and decrease by 50% or more with or without normalization of peripheral counts. Transfusion independence rate was calculated as the number of participants with neither RBC nor platelet transfusion for any period of 8 weeks after the initiation of treatment (or C1D1 visit date for participants randomized to BSC or randomization date for participants not treated) and up to treatment discontinuation (or 180 days for participants discontinuing the treatment within 6 months), while maintaining Hgb ≥8 g/dL and platelets ≥20×10^9/L divided by the total number of participants included in the efficacy analysis. The percentage of participants who achieved mCR and transfusion independence simultaneously in the same period were calculated for each group. Percentage of participants are rounded off to the single decimal point.
Time Frame: Up to approximately 46.6 months
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 277 | 140
percentage of participants | 5.8 | 2.9

4. Secondary Outcome: Survival Rate at 1 Year After Randomization
Description: One year survival rate was defined as the percentage of participants that survived at the end of the first year from randomization. Participants who did not have death in record were censored on the last date known to be alive. Percentage of participants are rounded off to the nearest whole number.
Time Frame: From randomization up to 12 months
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 277 | 140
percentage of participants | 39 [34 to 45] | 39 [30 to 47]

5. Secondary Outcome: Leukemia-free Survival
Description: Leukemia-free survival was defined as the number of days from randomization to the earliest date when participants have bone marrow (BM) or peripheral blood (PB) blasts ≥20%, conversion to acute myeloid leukemia (AML) or death of any cause. Participants with no events in leukemia-free survival were censored on the last date of BM or PB blasts assessment, whichever is later. Survival time will be estimated using the Kaplan-Meier method.
Time Frame: From randomization up to 46.6 months
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 277 | 140
days | 173.0 [135.0 to 206.0] | 181.0 [125.0 to 213.0]

6. Secondary Outcome: Number of Days Alive and Out of the Hospital (NDAOH)
Description: The date of each hospital admission and discharge was collected for each participant for up to 6 months, unless the participant died or withdrew consent prior to that time. Duration of each hospital stay in days was calculated as date of discharge minus date of admission. The NDAOH within first 6 month period was calculated as: NDAOH 6M=180 -total duration of all hospital stays within 180 days from the first treatment -number of death days before Day 180. For participants who were lost to follow-up within 6 months, the NDAOH was calculated conservatively assuming that the participant would have died the day after the last contact day.
Time Frame: Up to 6 months
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 277 | 140
days | 144.0 [0 to 180] | 149.5 [0 to 180]

7. Secondary Outcome: Disease Response (DR) Rate
Description: DR: Complete Response(CR), Partial Response(PR),Marrow Complete Response(mCR), and Hematological Improvement(HI) including HI with Erythroid (HI-E), HI with Neutrophil (HI-N), or HI with Platelet (HI-P) based on IWG 2006 criteria. CR: BM:≤5% myeloblasts, Peripheral blood: Hgb≥11g/dL, Platelets(PLTs)≥100x10^9/L, Neutrophils≥1.0x10^9/L, Blasts 0%. PR: All CR criteria if abnormal before treatment except BM blasts decreased ≥50% over pretreatment but still>5%, Cellularity, morphology not relevant. HI responses:1) HI-E: Hgb increase ≥1.5g/dL, Relevant reduction of RBC units transfusions by absolute ≥4 RBC transfusions/8 week(wk) compared with pretreatment transfusion number previous 8wk. Only RBC transfusions given for Hgb≤9.0g/dL. 2) HI-P: Absolute increase≥30x10^9/L starting>20x10^9/L PLTs; Increase from<20x10^9/L to>20x10^9/L and by≥100%. 3) HI-N: ≥100% increase, absolute increase>0.5x10^9/L.
Time Frame: Up to approximately 46.6 months
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment. Participants who had multiple responses of HI (HI-E, HI-N and HI-P) were counted only once while calculating the total HI value in both treatment groups. Percentage of participants are rounded off to the nearest single decimal point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 277 | 140
percentage of participants
  Complete Response (CR) | 1.4 [0.0 to 2.8] | 0.7 [0.0 to 2.1]
  Partial Response (PR) | 0 [0 to 0] | 0 [0 to 0]
  Marrow Complete Response (mCR) | 17.3 [12.9 to 21.8] | 8.6 [3.9 to 13.2]
  Hematological Improvement (HI) | 3.2 [1.2 to 5.3] | 5.7 [1.9 to 9.6]
  HI with Erythroid (HI-E) | 1.1 [0.0 to 2.2] | 2.1 [0.0 to 4.5]
  HI with Platelet (HI-P) | 1.8 [0.2 to 3.3] | 2.1 [0.0 to 4.5]
  HI with Neutrophil (HI-N) | 0.7 [0.0 to 1.7] | 2.1 [0.0 to 4.5]

8. Secondary Outcome: Duration of Complete Response (CR)
Description: Duration of complete response (in number of days) was calculated from the first time a CR was observed to the date of the earliest of the following three events: 1) relapse/disease progression, 2) start of alternative therapy (except Hematopoietic Cell Transplant [HCT]) or 3) death. In the absence of any event, the duration of CR was censored at the last available time point (BM assessment, PB assessment, or safety/long-term follow-up visit) at which an event was not observed. Duration of complete response was analysed using a Kaplan-Meier method for participants who achieved a CR during the study. CR: BM: ≤5% myeloblasts (all cell lines normal maturation), Peripheral blood: Hgb ≥11g/dL, PLTs ≥100x10^9/L, Neutrophils ≥1.0x10^9/L, Blasts 0%.
Time Frame: Up to approximately 46.6 months
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment. Overall number of participants analyzed are the number of participants with CR (responders) only.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 4 | 1
days | 198 [112.0 to 266.0] | 406 [NA to NA] — The upper and lower limit of 95% confidence interval was not estimable for a single participant.

9. Secondary Outcome: Time to First Response, Complete Response (CR) and Best Response
Description: Time to first response was the time(days) from randomization to first date when any response was achieved. Time to CR was the time(days) from randomization to first date when CR was achieved. Time to best response was the time(days) from randomization to first date when participant's best response (CR,PR,mCR or HI) was achieved. CR:BM:≤5% myeloblasts, Peripheral blood:Hgb≥11g/dL,PLTs≥100x10^9/L,Neutrophils≥1.0x10^9/L,Blasts 0%. PR: All CR criteria except BM blasts decreased≥50% over pretreatment but still >5%,Cellularity,morphology not relevant. mCR: Reduction of BM blasts to≤5%; decrease ≥50% with/without normalization of peripheral counts. HI responses:1)HI-E:Hgb increase≥1.5 g/dL, Relevant reduction of RBC units transfusions by absolute≥4 RBC transfusions/8wk compared with pretreatment transfusion number previous 8wk. 2)HI-P:Absolute increase≥30x10^9/L starting>20x10^9/L PLTs; Increase from≤20 to>20x10^9/L and by≥100% 3)HI-N:≥100% granulocyte increase, absolute increase>0.5x10^9/L.
Time Frame: From study Day 1 to the earliest date that a response was first documented (up to approximately 46.6 months)
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment. Overall number of participants analyzed are the number of participants with data available for analysis. 'Number Analyzed' indicates the number of participants with response.
Measure: Median (Full Range); unit: days
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 61 | 21
days
  Time to First Response (CR, PR, mCR, or HI) | 63.0 [28 to 323] | 67.0 [21 to 295]
  Time to CR: number analyzed (Participants) | 4 | 1
  Time to CR | 91.0 [56 to 106] | 266.0 [266.0 to 266.0]
  Time to Best Response (CR, PR, mCR, or HI) | 64.0 [28 to 469] | 77.0 [23 to 295]

10. Secondary Outcome: Number of Red Blood Cell (RBC) and Platelet Transfusions
Description: The total number of RBCs transfused or, separately, the total number of platelets transfused up to the 6-month time point for each participant was counted from the date of randomization to Day 180, the date of last contact, or date of death, whichever occurred earlier. One RBC or platelet transfusion was defined as one unit, and a single bag of RBCs or platelets was considered one unit. The mean total number of RBC or platelet units transfused per participant is presented.
Time Frame: Up to 6 months
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment.
Measure: Mean (Standard Deviation); unit: units of transfused RBC or platelet
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 277 | 140
units of transfused RBC or platelet
  RBC Transfusions | 18.9 (13.94) | 15.0 (13.53)
  Platelet Transfusions | 16.8 (18.64) | 12.1 (20.15)

11. Secondary Outcome: Change From Baseline in Health-related Quality of Life (QOL) By EuroQol 5-level 5-dimension (EQ-5D-5L) Summary Index
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L, first component is a descriptive system five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a second component visual analogue scale (VAS) that measures health state. Each dimension comprises 5 levels with corresponding numeric scores, where 1 indicates no problems, and 5 indicates extreme problems. The health status is converted to an index value using the country-specific weighted scoring algorithm for England. The summary index value for the England ranges from a worst score of -0.281 to a best score of 1. An increase in the EQ-5D-5L total score indicates improvement.
Time Frame: Baseline to Month 6
Population: The Efficacy Analysis Set included all participants randomly assigned to the study treatment. Overall number of participants analyzed are the number of participants with data available for analysis. 'Number Analyzed' indicates the number of participants with data available for analysis at the given timepoint. As pre-specified in the statistical analysis plan (SAP), the analysis included only the data collected for each participant during the first 6 months of study participation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 266 | 119
score on a scale
  Baseline | 0.8414 (0.1596) | 0.8404 (0.1587)
  Change from Baseline at Month 6: number analyzed (Participants) | 103 | 40
  Change from Baseline at Month 6 | -0.0386 (0.1466) | -0.0149 (0.1266)

12. Secondary Outcome: Change From Baseline in Health-related QOL: EuroQOL Visual Analogue Scale (EQ-VAS) Score
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. The second component, EQ VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine).
Time Frame: Baseline to Month 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 266 | 119
score on a scale
  Baseline | 71.24 (18.33) | 70.70 (18.32)
  Change from Baseline at Month 6: number analyzed (Participants) | 103 | 40
  Change from Baseline at Month 6 | -1.52 (16.39) | -2.43 (18.04)

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participants administered a drug; it does not necessarily have to have a causal relationship with this treatment. An SAE is defined any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization; results in persistent or significant disability; is congenital anomaly; is suspected transmission of any infectious agent via a medicinal product or is medically important. Treatment emergent AEs which are those with onset date on or after the date of the first dose of study drug on C1D1 until 30 days after the last dose of study treatment, or the start of an alternative anticancer treatment, whichever occurs first.
Time Frame: From first dose through end of study (up to approximately 46.6 months)
Population: The Safety Analysis Set included all participants randomly assigned to study treatment who received any amount of study treatment or any component of a multi-dose study treatment regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 270 | 122
Participants
  TEAE | 268 | 113
  SAE | 216 | 65

14. Secondary Outcome: 30-day and 60-day All-cause Mortality
Description: Number of deaths, regardless of cause, within 30 or 60 days from the first study dose divided by the total number of participants included in the Safety Analysis Set. Participants who died within 30 days were also included in the 60-day mortality calculations.
Time Frame: From first dose until 60 days after study treatment initiation
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Guadecitabine | Treatment Choice
Number analyzed (Participants) | 270 | 122
Participants
  Within 30 Days | 16 | 6
  Within 60 days | 35 | 13

ADVERSE EVENTS:
Time Frame: From first dose through end of study (up to approximately 46.6 months)
Description: All-cause mortality:The Efficacy Analysis Set included all participants randomly assigned to study treatment.
  Serious and other adverse events:The Safety Analysis Set included all participants randomly assigned to study treatment who received any amount of study treatment or any component of a multi-dose study treatment regimen.
  As pre-specified in the protocol, participants were grouped, and data was collected according to treatment received (Guadecitabine/Treatment Choice)for adverse events.
Arm/Group | Guadecitabine | Treatment Choice
All-Cause Mortality (participants affected / at risk) | 237/277 | 122/140
Serious Adverse Events (participants affected / at risk) | 216/270 | 65/122
Other Adverse Events (participants affected / at risk) | 266/270 | 107/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Guadecitabine (N=270) | Treatment Choice (N=122)
Febrile Neutropenia (Blood and lymphatic system disorders) | 80 | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 2
Anaemia (Blood and lymphatic system disorders) | 7 | 2
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Leukostasis Syndrome (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Splenic Infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 6 | 1
Cardiac Failure (Cardiac disorders) | 4 | 2
Cardiac Failure Congestive (Cardiac disorders) | 3 | 0
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0
Angina Pectoris (Cardiac disorders) | 2 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 1
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0
Gastrointestinal Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Chronic Gastritis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Enterovesical Fistula (Gastrointestinal disorders) | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Vascular Malformation Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Megacolon (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Retroperitoneal Haematoma (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 2
General Physical Health Deterioration (General disorders) | 3 | 3
Multiple Organ Dysfunction Syndrome (General disorders) | 2 | 0
Chest Pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 2
Malaise (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 1
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 72 | 17
Sepsis (Infections and infestations) | 26 | 4
Septic Shock (Infections and infestations) | 16 | 2
Cellulitis (Infections and infestations) | 14 | 2
Bacteraemia (Infections and infestations) | 11 | 1
Urinary Tract Infection (Infections and infestations) | 5 | 3
Bronchopulmonary Aspergillosis (Infections and infestations) | 4 | 0
Infection (Infections and infestations) | 4 | 1
Urosepsis (Infections and infestations) | 4 | 0
Anal Abscess (Infections and infestations) | 3 | 0
Device Related Infection (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis Orbital (Infections and infestations) | 2 | 0
Chronic Sinusitis (Infections and infestations) | 2 | 0
Corynebacterium Infection (Infections and infestations) | 2 | 0
Pseudomonal Bacteraemia (Infections and infestations) | 2 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 2 | 0
Subcutaneous Abscess (Infections and infestations) | 2 | 0
Abscess Jaw (Infections and infestations) | 1 | 0
Anorectal Infection (Infections and infestations) | 1 | 0
Brain Abscess (Infections and infestations) | 1 | 1
Clostridial Infection (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Corona Virus Infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Endophthalmitis (Infections and infestations) | 1 | 0
Enterococcal Infection (Infections and infestations) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Fungal Infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Haematoma Infection (Infections and infestations) | 1 | 0
Herpes Virus Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Metapneumovirus Infection (Infections and infestations) | 1 | 0
Mucormycosis (Infections and infestations) | 1 | 0
Necrotising Fasciitis (Infections and infestations) | 1 | 0
Necrotising Soft Tissue Infection (Infections and infestations) | 1 | 0
Otitis Media Acute (Infections and infestations) | 1 | 0
Periorbital Cellulitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumococcal Sepsis (Infections and infestations) | 1 | 0
Pseudomembranous Colitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 1
Sinusitis Fungal (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0
Streptococcal Bacteraemia (Infections and infestations) | 1 | 0
Streptococcal Endocarditis (Infections and infestations) | 1 | 0
Streptococcal Infection (Infections and infestations) | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection Staphylococcal (Infections and infestations) | 1 | 0
Vulval Cellulitis (Infections and infestations) | 1 | 0
Wound Abscess (Infections and infestations) | 1 | 0
Candida Infection (Infections and infestations) | 0 | 1
Clostridium Bacteraemia (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Nocardiosis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Acute Haemolytic Transfusion Reaction (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 2
C-Reactive Protein Increased (Investigations) | 1 | 0
General Physical Condition Abnormal (Investigations) | 1 | 0
Troponin Increased (Investigations) | 1 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Fistula Inflammation (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central Nervous System Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 2 | 2
Central Nervous System Haemorrhage (Nervous system disorders) | 1 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Intracranial Haematoma (Nervous system disorders) | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Organic Brain Syndrome (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Tract Pain (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1/194 | 0/96 — Number of participants at risk are based on the male population.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 2
Internal Haemorrhage (Vascular disorders) | 1 | 0
Shock Haemorrhagic (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Guadecitabine (N=270) | Treatment Choice (N=122)
Anaemia (Blood and lymphatic system disorders) | 63 | 22
Febrile Neutropenia (Blood and lymphatic system disorders) | 38 | 6
Leukopenia (Blood and lymphatic system disorders) | 32 | 12
Neutropenia (Blood and lymphatic system disorders) | 92 | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 84 | 25
Abdominal Pain (Gastrointestinal disorders) | 27 | 6
Constipation (Gastrointestinal disorders) | 62 | 12
Diarrhoea (Gastrointestinal disorders) | 60 | 20
Haemorrhoids (Gastrointestinal disorders) | 16 | 4
Nausea (Gastrointestinal disorders) | 43 | 15
Stomatitis (Gastrointestinal disorders) | 38 | 7
Vomiting (Gastrointestinal disorders) | 29 | 7
Asthenia (General disorders) | 53 | 12
Fatigue (General disorders) | 59 | 11
Injection Site Reaction (General disorders) | 46 | 1
Oedema (General disorders) | 14 | 9
Oedema Peripheral (General disorders) | 42 | 14
Pyrexia (General disorders) | 60 | 24
Cellulitis (Infections and infestations) | 22 | 4
Nasopharyngitis (Infections and infestations) | 10 | 7
Pneumonia (Infections and infestations) | 40 | 8
Upper Respiratory Tract Infection (Infections and infestations) | 16 | 7
Urinary Tract Infection (Infections and infestations) | 13 | 7
Contusion (Injury, poisoning and procedural complications) | 24 | 8
Fall (Injury, poisoning and procedural complications) | 17 | 5
Transfusion Reaction (Injury, poisoning and procedural complications) | 17 | 3
Alanine Aminotransferase Increased (Investigations) | 13 | 8
Aspartate Aminotransferase Increased (Investigations) | 10 | 8
Blood Creatinine Increased (Investigations) | 14 | 5
Weight Decreased (Investigations) | 22 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 49 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 45 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 33 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 17 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 15 | 7
Dizziness (Nervous system disorders) | 34 | 8
Headache (Nervous system disorders) | 34 | 9
Insomnia (Psychiatric disorders) | 31 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 44 | 21
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14 | 3
Erythema (Skin and subcutaneous tissue disorders) | 14 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 24 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 2
Rash (Skin and subcutaneous tissue disorders) | 27 | 7
Haematoma (Vascular disorders) | 15 | 5
Hypotension (Vascular disorders) | 17 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT02907359/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT02907359/SAP_001.pdf